CLINICAL TRIAL: NCT03308097
Title: A Mobile Intervention to Improve Uptake of PrEP for Southern Black MSM
Acronym: MobilePrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH111342 (NIH)
Record Dates: First submitted 2017-10-02; First posted 2017-10-12 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-01

CONDITIONS: Hiv
Keywords: PrEP; Uptake; MSM; Black
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP Mobile Messaging Intervention (Experimental): Participants from the STI/HIV testing clinic will receive Enhanced Standard of Care (described below) plus texted messages with the intervention content and follow-up questions over the next 4 weeks on their cell phones. Participants will receive approximately 8-16 interactive text messages with links to web content. Texts will be sent twice a week over the next 4 weeks. Participants will return for 2 more appointments over the next couple of months to fill out questionnaires.
  Interventions: Behavioral: PrEP Mobile Messaging Intervention
- Enhanced Standard of Care (Active Comparator): As part of the enhanced standard of care, participants seen in the STI/HIV testing clinic are given feedback regarding PrEP eligibility and current risk behaviors. Participants are also given an informational handout about PrEP, shown a brief video, and given contact information for the PrEP Clinic Care Coordinator. Participants will return for 2 more visits over the next couple months to fill out questionnaires.
  Interventions: Behavioral: Enhanced Standard of Care

INTERVENTIONS:
Behavioral: PrEP Mobile Messaging Intervention — See group description
  Arms: PrEP Mobile Messaging Intervention
Behavioral: Enhanced Standard of Care — See group description
  Arms: Enhanced Standard of Care

SUMMARY:
This study will develop and test an interactive mobile messaging intervention to improve engagement in care related to Pre-exposure Prophylaxis (PrEP) and decrease HIV risk behaviors for Black men who have sex with men living in the Southern U.S. The mobile messaging intervention will include interactive text messaging and free, publicly available links to websites and YouTube videos. During the intervention participants will gain information about their health, improve motivation for engagement in PrEP related care, and build skills for healthy behaviors. Participants will also receive intervention materials to help decrease frequent barriers to care. If the intervention is found to be effective, it can be tested in a larger study and then disseminated.

DETAILED DESCRIPTION:
The uptake of Pre-Exposure Prophylaxis (PrEP) has been slow for young Black men who have sex with men (BMSM) living in the Southern United States. This is a significant issue because eight of the ten states with the highest rates of new HIV infections are located in the South. Jackson, Mississippi (MS) (the site of this project) has the second highest AIDS diagnosis rate in the nation, and the highest rate of HIV infection for young urban Black men who have sex with men. This study will develop and test an engaging, interactive, and cost effective mobile messaging intervention to improve linkage to PrEP care for BMSM (18-35 yrs) living in Jackson, MS. BMSM eligible for PrEP, receiving care at the University of Mississippi Medical Center sexually-transmitted infections (STI)/HIV testing clinics, will be texted interactive links to publicly available, online content about PrEP and HIV prevention. Links will be sent to PrEP eligible BMSM by 8-16 interactive text messages over 4 weeks. The material used in the intervention will be consistent with the Information Motivation Behavior (IMB) Model and will address cultural and structural barriers to initiating PrEP care. A small randomized controlled study among 66 new participants in the clinics will examine the preliminary efficacy of the intervention compared to enhanced standard of care on attendance at a PrEP Services Appointment (the first step in initiating PrEP care). It is hypothesized that, compared to BMSM receiving enhanced standard of care, BMSM receiving the PrEP Mobile Messaging Intervention will show greater attendance at a PrEP Services Appointment and decreased HIV risk behavior at 4 and 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Black MSM
* Eligible for PrEP
* Visit STI/HIV testing clinics at University of Mississippi Medical Center
* Able to give consent/assent and not impaired by cognitive or medical limitations as per clinical assessment

Exclusion Criteria:

- Involved in another PrEP or HIV prevention related study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Study only open to self-identifying male participants.
Enrollment: 70 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry K. Brown, M.D., Principal Investigator — Rhode Island Hospital; Laura Whiteley, M.D., Principal Investigator — Rhode Island Hospital; Leandro Mena, M.D., Study Director — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Derived] Rouffiac AE, Whiteley L, Brown L, Mena L, Craker L, Healy M, Haubrick K. A Mobile Intervention to Improve Uptake of Pre-Exposure Prophylaxis for Southern Black Men Who Have Sex With Men: Protocol for Intervention Development and Pilot Randomized Controlled Trial. JMIR Res Protoc. 2020 Feb 20;9(2):e15781. doi: 10.2196/15781. PMID 32130196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 70 individuals completed consent are were enrolled.
Pre-assignment Details: Of the 70 enrolled participants, 68 completed baseline assessment- 1 did not return to the clinic to complete baseline and another seroconverted and was no longer eligible.
  Of the 68 participants who completed baseline, 65 were randomized- 2 were confirmed HIV+ and no longer eligible, and 1 previously worked at UMMC and was removed from the study.
Period: Overall Study
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
Started | 33 | 32
Completed | 31 | 31
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (4.8) | 23.6 (4.8) | 23.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 33 | 32 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 30 | 31 | 61
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 28 | 56
  White | 0 | 0 | 0
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 1 | 3
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 0 | 1 | 1
  Homosexual | 19 | 24 | 43
  Bisexual | 10 | 5 | 15
  Asexual | 1 | 0 | 1
  Undecided | 0 | 1 | 1
  Unknown/Not reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of PrEP Services Appointments Attended-Full Sample
Description: With participant consent, staff at the STI/HIV testing clinic will abstract from the electronic medical record any PrEP Services Appointment, and any PrEP related care.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: visits attended
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 31 | 31
visits attended | 0.58 (0.72) | 0.55 (0.68)

2. Primary Outcome: Number of PrEP Services Appointments Attended- Restricted Sample
Description: With participant consent, staff at the STI/HIV testing clinic will abstract from the electronic medical record any PrEP Services Appointment, and any PrEP related care.
  Restricted Sample is only those who did not receive a PrEP prescription the same day as enrollment.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: visits attended
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 27 | 26
visits attended | 0.56 (0.75) | 0.50 (0.65)

3. Primary Outcome: Number of Participants Who Received a PrEP Prescription-Full Sample
Description: Staff at the testing clinic will abstract any prescription written for PrEP at 16 weeks for the participant.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 31 | 31
Participants
  Did not receive PrEP Prescription | 16 | 17
  Received PrEP Prescription | 15 | 14

4. Primary Outcome: Number of Participants Who Received a PrEP Prescription-Restricted Sample
Description: Staff at the testing clinic will abstract any prescription written for PrEP at 16 weeks for the participant.
  Restricted sample is those who did not receive a PrEP prescription the same day as enrollment.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 27 | 26
Participants
  Did not receive PrEP Prescription | 16 | 16
  Received PrEP Prescription | 11 | 10

5. Secondary Outcome: Change in PrEP Knowledge-Full Sample
Description: Change in participants score on the PrEP Knowledge Questionnaire between baseline and 16 weeks follow-up. Scores can range from 0-3, with higher scores indicating greater PrEP knowledge.
Time Frame: Baseline, 16 weeks
Population: Missing data accounts for the discrepancy in the analytic sample for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 24 | 28
score on a scale | 0.50 (0.83) | 1.00 (1.15)

6. Secondary Outcome: Change in PrEP Knowledge-Restricted Sample
Description: Change in participants score on the PrEP Knowledge Questionnaire between baseline and 16 weeks follow-up. Scores can range from 0-3, with higher scores indicating greater PrEP knowledge.
  Restricted sample is those who did not receive a PrEP prescription the same day as enrollment.
Time Frame: Baseline, 16 weeks
Population: Missing data accounts for the discrepancy in the analytic sample for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 22 | 23
score on a scale | 0.55 (0.86) | 0.83 (1.15)

7. Secondary Outcome: Change in Social Motivational Readiness for PrEP Care-Full Sample
Description: Change in participants' score on the IMB PrEP Motivation Scale (to assess personal and social motivations for PrEP use) from baseline to16 weeks follow-up. Scores can range from 8 - 32, with higher scores indicating greater motivation.
Time Frame: Baseline, 16 weeks
Population: Missing data accounts for the discrepancy in the analytic sample for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 19 | 24
units on a scale | -1.00 (3.59) | 0.29 (4.46)

8. Secondary Outcome: Change in Social Motivational Readiness for PrEP Care-Restricted Sample
Description: Change in participants' score on the IMB PrEP Motivation Scale (to assess personal and social motivations for PrEP use) from baseline to16 weeks follow-up. Scores can range from 8 - 32, with higher scores indicating greater motivation.
  Restricted sample is those who did not receive a PrEP prescription the same day as enrollment.
Time Frame: Baseline, 16 weeks
Population: Missing data accounts for the discrepancy in the analytic sample for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 17 | 19
units on a scale | -1.35 (3.48) | 0.47 (4.72)

9. Secondary Outcome: Change in PrEP Self-efficacy-Full Sample
Description: Change in participants' score on the IMB PrEP Behavioral Skills Scale between baseline and 16 weeks, which assesses self-efficacy for taking PrEP as prescribed and assesses self-efficacy for PrEP related medical appointments. Scores can range from 7 - 28, with higher scores indicating greater self-efficacy.
Time Frame: Baseline, 16 weeks
Population: Missing data accounts for the discrepancy in the analytic sample for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 15 | 19
score on a scale | -0.33 (3.11) | -0.37 (2.91)

10. Secondary Outcome: Change in PrEP Self-efficacy-Restricted Sample
Description: Change in participants' score on the IMB PrEP Behavioral Skills Scale between baseline and 16 weeks, which assesses self-efficacy for taking PrEP as prescribed and assesses self-efficacy for PrEP related medical appointments. Scores can range from 7 - 28, with higher scores indicating greater self-efficacy.
  Restricted sample is those who did not receive a PrEP prescription the same day as enrollment.
Time Frame: Baseline, 16 weeks
Population: Missing data accounts for the discrepancy in the analytic sample for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 14 | 15
score on a scale | -0.36 (3.23) | -0.20 (3.21)

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events over the duration of the study (4 months).
Arm/Group | PrEP Mobile Messaging Intervention | Enhanced Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT03308097/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-11-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT03308097/Prot_SAP_001.pdf